CLINICAL TRIAL: NCT06949722
Title: Redirecting Poor Sleep Drivers of Early Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Michael W.L. Chee, Professor, National University of Singapore
Other Study IDs: RESET-Sleep
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Sleep; Cardiovascular Risk Factors
Keywords: Sleep; Cardiovascular disease; Wearables; Cardiovascular risk; Objective sleep tracking
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from RESET: Interested participants will be drawn from the RESET cohort which includes South-East Asians aged 40-70 years with no prior manifest atherosclerotic cardiovascular disease.

SUMMARY:
Sleep health is a critical component of cardiovascular well-being, and poor sleep has been linked with increased risk for all-cause mortality including cardiovascular disease (CVD). Moreover, many individuals within a population may have underlying, subclinical cardiovascular conditions, such as hypertension and arterial stiffness, and these may risk progressing to advanced CVD when coupled with inadequate sleep duration and quality. Given that Singapore ranks as the third most sleep-deprived city globally, understanding the relationship between sleep health and the prevalence and progression of CVD becomes increasingly important for population health. In addition, depression and psychological stress could also lead to poorer cardiovascular health by increasing blood cholesterol, blood sugar and blood pressure, and could also be directly related to or arise as a result of poor sleep. The aim of the current study is to track sleep and mental health using a combination of objective sleep tracking (Oura ring) and smartphone-based questionnaires (EMA), and examine their associations with detailed cardiovascular health data collected by the project RESET (Redirecting Immune, Lipid and Metabolic Drivers of Early Cardiovascular Disease).

DETAILED DESCRIPTION:
Sleep health is a critical component of cardiovascular well-being, and poor sleep has been linked with increased risk for all-cause mortality including cardiovascular disease (CVD). Previous research suggested that inadequate duration and quality of sleep may increase the risk for developing cardiovascular disease. Moreover, many individuals within a population may have underlying, subclinical cardiovascular conditions, such as hypertension and arterial stiffness, and these may risk progressing to advanced CVD when coupled with poor sleep. Given that Singapore ranks as the third most sleep-deprived city globally, understanding the relationship between sleep health and the prevalence and progression of CVD becomes increasingly important for population health. In addition, depression and psychological stress could also lead to poorer cardiovascular health. by increasing blood cholesterol, blood sugar and blood pressure, and could also be directly related to or arise as a result of poor sleep. Therefore, it is essential to assess the relationship between CVD progression and sleep as a multidimensional construct with overlapping components, including duration, timing, regularity, and efficiency, using objectively collected data over multiple days.

Through the combination of objective sleep tracking through wearables with health assessments conducted in the RESET study (registered with ClinicalTrials.gov under NCT06211868), we will gain valuable insights into these dimensions of poor sleep and wellbeing factors that are associated with poor cardiovascular health.

The investigators aim to examine following questions using a combination of objective sleep tracking (Oura ring), smartphone-based questionnaires (EMA) and detailed health data collected by the RESET study.

1. How are sleep patterns, in terms of duration, timing, efficiency and regularity, associated with cardiovascular health outcomes and disease risk, at baseline and follow-up ?
2. How are sleep patterns, in terms of duration, timing, efficiency and regularity, associated with vascular aging patterns?
3. How are patterns of subjective wellbeing related to cardiovascular health, at baseline and follow-up ?
4. Do sleep and subjective wellbeing measures relate on a day to day basis?

The investigators hypothesize that inadequate sleep duration, timing, and regularity will be associated with increased cardiovascular risk at baseline and follow-up. Individuals with irregular sleep duration and timing are expected to demonstrate higher arterial stiffness and profiles indicative of early vascular aging. Additionally, participants reporting poor subjective well-being are anticipated to experience poorer sleep quality, which will further associate with increased cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Willing to wear a ring
* Have any of the following conditions:

  * High blood pressure
  * High cholesterol
  * Fatty liver
  * Family history of heart diseases or stroke.
  * Obesity

Exclusion Criteria:

* Prior history of heart attack or stroke or balloon angioplasty/stent placement
* Restricted peripheral circulation (e.g., Raynaud's disease)
* Pacemakers

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: South-East Asian population aged 40-70 years with no prior manifest atherosclerotic cardiovascular disease (ACSVD).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sleep time | Across the 2 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Onset Time, Wake Time, on Workday (weekday) and Free Day (Weekend / vacation) will be recorded for nocturnal sleep and naps.
Sleep duration | Across the 2 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Duration on Workday (weekday) and Free Day (Weekend / vacation) will be recorded for nocturnal sleep and naps.
Wake after sleep onset | Across the 2 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Wake after Sleep Onset on Workday (weekday) and Free Day (Weekend / vacation) will be recorded.
Sleep regularity | Across the 2 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Regularity (computed via Std Deviation and Sleep Regularity Index; evaluated over 4 weeks minimally) will be recorded.
Well-being | Across the 2 year study
  Participants input ratings about a rotating set of questions concerning wellbeing daily through a smartphone based app (Z4IP) that has been used in prior studies. This daily assessment can be done anytime between 8pm and 12am each day. Higher scores represent higher levels of well-being.
Major adverse cardiovascular event | Across the 2 year study
  Composite of cardiac death, non-fatal myocardial infarction, resuscitated cardiac arrest, non-fatal ischemic stroke, congestive heart failure, coronary revascularization
Arterial stiffness | Across the 2 year study
  Pulse wave velocity and arterial stiffness measurements will be recorded using applanation tonometry
Vascular age | Across the 2 year study
  Vascular age is calculated using arterial stiffness and traditional cardiovascular risk factors to infer about vascular health.

SECONDARY OUTCOMES:
Predicted vascular age | Across the 2 year study
  Vascular age will be predicted using PPG data and machine learning approaches.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No